CLINICAL TRIAL: NCT01653561
Title: A Multi-institutional, Open-label, Single Arm Study of Apatinib in Non-triple-negative Metastatic Breast Cancer
Brief Title: A Study of Apatinib in Non-triple-negative Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xichun Hu, Deputy director of department of medical oncology, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fudan BR2012-08
Record Dates: First submitted 2012-07-10; First posted 2012-07-31 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-08

CONDITIONS: Breast Neoplasms
Keywords: Metastatic breast cancer; Apatinib; non-triple-negative
MeSH Terms: conditions — Breast Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Apatinib (Experimental): Apatinib 500mg/d
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — The starting dose of apatinib will be 500mg/d. Two dose reductions will be allowed to 375 and then 250 mg/d.

SUMMARY:
The hypothesis of this clinical research study is to discover if the study drug apatinib can shrink or slow the growth of pretreated non-triple-negative metastatic breast cancer.

DETAILED DESCRIPTION:
Apatinib is a tyrosine kinase inhibitor targeting vascular endothelial growth factor receptor (VEGFR), and its anti-angiogenesis effect has been viewed in preclinical tests. The investigators' phase I study has shown that the drug's toxicity is manageable and the maximum tolerable daily dose is 850 mg. The hypothesis of this clinical research study is to discover if the study drug apatinib can shrink or slow the growth of non-triple-negative breast cancer. The safety of apatinib will also be studied. Patients physical state, symptoms, changes in the size of the tumor, and laboratory findings obtained while on-study will help the research team decide if apatinib is safe and effective in pretreated non-triple-negative metastatic breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

●≥ 18 and ≤ 70 years of age.

* ECOG performance status of 0-1.
* Metastatic breast cancer, confirmed by histological analysis.
* Have experienced at least 1 and at most 4 regimens, and failed from the last chemotherapy regimen. Pretreated anthracycline, taxanes and capecitabine (any rational reason for no use of capecitabine is acceptable) are mandatory.
* Women diagnosed with human epidermal growth factor receptor positive (HER2+) should have failed for at least 1 anti-HER2 therapy (any rational reason for no use of anti-HER2 therapy is acceptable). HER2+ is defined as +++ staining on immunohistochemistry or FISH/CISH positive for gene amplification.
* Women diagnosed with HR+ should have failed for at least 1 hormonal therapy.
* Have failed for at least one chemotherapy regimen, but at most three regimens(including adjuvant and neo-adjuvant setting).
* Duration from the last therapy (chemotherapy, radiotherapy, target therapy and operation) is more than 4 weeks (Duration for nitroso or mitomycin is 6 weeks).
* Have at least one extracranial measurable site of disease according to RECIST 1.0 criteria that has not been previously irradiated.
* Life expectancy of more than 3 months.
* Negative serum or urine pregnancy test taken in all women within 7 days before inclusion. Sexually active women of childbearing potential must use a medically acceptable form of contraception from the beginning of the study to 8 weeks after the last dose of the investigated drug.
* Written informed consent prior to study specific screening procedures.

Exclusion Criteria:

* Triple-negative breast cancer (ER-, PR- and HER2-. HER2- is defined as 0 or 1+ staining on immunohistochemistry or FISH/CISH negative for gene amplification. )
* Pregnant or lactating women.
* Less than 4 weeks from the last clinical trial.
* Uncontrolled hypertension with mono-drug therapy (>140/90 mm Hg)；ischemia of the myocardium （≥ grade 2） or myocardial infarction；arrhythmia（≥ grade 2, QTcF > 470ms for female patients） or New York Heart Association Class III/IV
* Any factors that influence the usage of oral administration.
* The cumulative doses of doxorubicin and epirubicin before inclusion have surpassed 300 mg/m2 and 600 mg/m2, respectively.
* Duration from the last therapy (chemotherapy, radiotherapy, target therapy and operation) is less than 4 weeks (Duration for nitroso or mitomycin is less than 6 weeks).
* Confirmed brain metastasis.
* Inadequate hepatic, renal, heart, and hematologic functions (hemoglobin <90g/L, neutrophils < 1.5×10^9/L, platelets < 80×10^9/L , ALT > 2.5 x upper limit of normal (ULN)(5x for liver metastasis), AST > 2.5 x ULN (5x for liver metastasis), serum bilirubin > 1.5 x ULN, serum creatine > 1.0 x ULN, creatinine clearance rate ≤ 50ml/min, LVEF < lower limit of normal (LLN).
* Abnormal coagulative function, inclined to bleeding or is receiving thrombolytictherapy or anticoagulation.
* History of arterial/venous embolic events (such as cerebrovascular accident, TIA, deep vein thrombus,and pulmonary embolism)
* Unhealed wound (> 30 days) or bone fracture.
* Urine protein ≥++ and confirmed >1.0 g by the 24h quantity.
* Previous or present history of pulmonary fibrosis,interstitial pneumonia,pneumoconiosis,radiation pneumonitis,drug-related pneumonitis or greatly-impaired pulmonary function.
* Disability of serious uncontrolled intercurrence infection.
* Abuse of alcohol or drugs.
* Have received prior treatment with a VEGFR, PDGFR or s-SRC TKI (Bevacizumab is permitted).
* Acquired or inherent immunodeficiency； HIV infection； organ transplantation history.
* The active HBV or HCV infection or HBV DNA ≥10^4/ml.
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix.
* Presence of serious harm to subjects or complication to hinder the completion of the study judged by investigators

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
PFS(Progression free survival) | 8 Weeks

SECONDARY OUTCOMES:
ORR (Objective response rate) | 8 Weeks
CBR(Clinical benefit rate) | 8 Weeks
OS (Overall survival) | 8 Weeks
QoL (Quality of life) | 8 Weeks
Toxicity (Number of adverse events) | 8 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xi-Chun Hu, Doctor, Principal Investigator — Fudan Univeristy Cancer Hospital
Locations (2):
- China (2):
  - Fudan University Cancer Hospital, Shanghai, Shanghai Municipality
  - Fudan University Cancer Hospital, Shanghai

REFERENCES:
- [Derived] Hu X, Cao J, Hu W, Wu C, Pan Y, Cai L, Tong Z, Wang S, Li J, Wang Z, Wang B, Chen X, Yu H. Multicenter phase II study of apatinib in non-triple-negative metastatic breast cancer. BMC Cancer. 2014 Nov 7;14:820. doi: 10.1186/1471-2407-14-820. PMID 25376790
- [Derived] Fan M, Zhang J, Wang Z, Wang B, Zhang Q, Zheng C, Li T, Ni C, Wu Z, Shao Z, Hu X. Phosphorylated VEGFR2 and hypertension: potential biomarkers to indicate VEGF-dependency of advanced breast cancer in anti-angiogenic therapy. Breast Cancer Res Treat. 2014 Jan;143(1):141-51. doi: 10.1007/s10549-013-2793-6. Epub 2013 Dec 1. PMID 24292957